CLINICAL TRIAL: NCT04490408
Title: Long Surgical Bypass Versus Hybrid Approaches for Management of Critical Limb Ischemia
Brief Title: Surgical Bypass Versus Hybrid Approaches for Critical Limb Ischemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Egyptian Biomedical Research Network (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EBRN71
Record Dates: First submitted 2020-07-24; First posted 2020-07-29 (Actual); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Critical Lower Limb Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- long surgical bypass (Active Comparator): long surgical bypass for multilevel lower limb ischemia
  Interventions: Procedure: long surgical bypass
- Hybrid approach (Experimental): surgical bypass and endovascular treatment for multilevel lower limb ischemia
  Interventions: Procedure: Hybrid approach

INTERVENTIONS:
Procedure: long surgical bypass — long surgical bypass and hybrid approaches in patients with multilevel critical lower limb ischemia.
  Arms: long surgical bypass
Procedure: Hybrid approach — Hybrid approach including bypass and endovascular revascularization
  Arms: Hybrid approach

SUMMARY:
The present randomized study proposed to compare the immediate postoperative and 2-year clinical outcomes of long surgical bypass and hybrid approaches in patients with multilevel critical lower limb ischemia.

ELIGIBILITY:
Inclusion Criteria:

* TASC II type D femoropopliteal lesions with intact ipsilateral femoral pulse.
* Fontaine classification stage IV (gangrene or necrosis).
* Rutherford grade III and IV category 5 and 6 with salvageable foot

Exclusion Criteria:

* heart failure
* liver failure
* renal impairment

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2014-09-20 (Actual); Primary Completion 2019-04-17 (Actual); Study Completion 2019-04-17 (Actual)

PRIMARY OUTCOMES:
Late occlusion | 2 years
  Late occlusion of the affected vessels

IPD SHARING:
Plan to Share IPD: No